CLINICAL TRIAL: NCT03773510
Title: Time to Secondary Resistance to Trabectedin After Interruption Versus Continuation in Responding Patients With Liposarcoma, Leiomyosarcoma and Synovial Sarcoma
Brief Title: Study on Leiomyosarcoma, Liposarcomas and Synovial Sarcoma With Trabectedin
Acronym: TRADITIONS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Not approved by the coordinating Ethical Committee
Sponsor: Italian Sarcoma Group (Network)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISG TRADITIONS
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Leiomyosarcoma; Liposarcoma; Synovial Sarcoma
Keywords: trabectedin; soft tissue sarcoma
MeSH Terms: conditions — Leiomyosarcoma; Liposarcoma; Sarcoma, Synovial; Sarcoma

STUDY DESIGN:
Intervention Model Description: Randomized, open-label , two arm study All the patients who will complete 6 cycles of treatment without disease progression will be be randomized to continue Trabectedin versus "treatment interruption" followed by re-challenge at progression. Patients randomized to discontinue treatment will be candidate to other 6 cycles of treatment and if they do not progress, to another interruption. The treatment will be resumed again at progression for other 6 cycles and this scheme of treatment will be proposed until progression under Trabectedin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trabectedin continuation (Active Comparator): All the patients who will complete 6 cycles of trabectedin without disease progression, will continue trabectedin until progressive disease, unacceptable toxicity, patient or investigator decision
  Interventions: Drug: Trabectedin continuation
- Trabectedin discontinuation (Experimental): All the patients who will complete 6 cycles of trabectedin without disease progression , will discontinue trabectedin.
  The treatment will be resumed again at progression for other 6 cycles and this scheme of treatment will be proposed until progression under trabectedin.
  Interventions: Drug: Trabectedin discontinuation

INTERVENTIONS:
Drug: Trabectedin discontinuation — Patients who did not progressed after 6 cycles of trabectedin will stop the treatment and resume drug in case of progression for other 6 cycles.
  The treatment will be resumed again at progression for other 6 cycles and this scheme of treatment will be proposed until progression under trabectedin.
  Other Names: Treatment discontinuation
  Arms: Trabectedin discontinuation
Drug: Trabectedin continuation — Patients who did not progressed after 6 cycles of trabectedin will continue the treatment until Progressive Disease or unacceptable toxicity
  Other Names: Treatment continuation
  Arms: Trabectedin continuation

SUMMARY:
Two arm, randomized, open-label study, to determine the best time to secondary resistance between responding patients who discontinue treatment and resumed Trabectedin at the time of progression versus patients who continued treatment until progression. T

DETAILED DESCRIPTION:
This is an Italian, multicenter, randomized, open-label , two arm, study, to determine the best time to secondary resistance between responding patients who discontinue treatment and resumed Trabectedin at the time of progression versus patients who continued treatment until progression. The aim is to evaluate the best clinical practice for responding patients as Trabectedin has an acceptable safety profile with no evidence of cumulative toxicity.

After signing informed consent and being assessed for eligibility criteria , eligible patients will start the trabectedin treatment.

All the patients who will complete 6 cycles of treatment without disease progression will be be randomized to continue Trabectedin versus "treatment interruption" followed by re-challenge at progression. Patients randomized to discontinue treatment will be candidate to other 6 cycles of treatment and if they do not progress, to another interruption. The treatment will be resumed again at progression for other 6 cycles and this scheme of treatment will be proposed until progression under Trabectedin.

The study will be conducted in Italy in approximately 12 centers, in order to recruit 330 evaluable patients over a 4 year period. The follow-up will last approximately 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or legal representative must be able to read and understand the informed consent form and must have been willing to give written informed consent and any locally required authorization before any study-specific procedures, including screening evaluations, sampling, and analyses
2. Diagnosis of well differentiated/dedifferentiated liposarcoma, mixoid round cell liposarcoma, leiomyosarcoma or synovial sarcoma
3. Persistent or locally relapsed and/or metastatic disease
4. Pathology specimens available for centralized review (central review is not mandatory prior to start the treatment, but within a month from screening, tumor sample must be sent to central pathology reviewer for a retrospective diagnosis confirmation).
5. Age ≥ 18 years
6. Adequate bone marrow function
7. Adequate organ function,
8. Eastern Cooperative Oncology Group Performance Status ≤ 2
9. One or more previous systemic treatments with anthracyclines with or without ifosfamide (unless one or both are clinically contraindicated)
10. Measurable disease. Patient who received radiotherapy within 3 weeks form the treatment start, can be included as long there is a measurable lesion outside of the irradiation field
11. A minimum of 3 weeks since any previous chemotherapy treatment
12. Recovery from toxic effects of prior therapies to (Grade 1 or lower)
13. Female patients of child-bearing potential must have negative pregnancy test within 7 days before initiation each cycle of chemotherapy. Post-menopausal women must be amenorrhoeic for at least 12 months to be considered of non-childbearing potential. Male and female patients of reproductive potential must agree to employ an effective method of birth control throughout the study.

Exclusion Criteria:

1. Pregnant or breast-feeding women
2. Prior exposure to Trabectedin
3. Peripheral neuropathy, Grade 2 or higher
4. History of other malignancies (except basal cell carcinoma or cervical carcinoma in situ, adequately treated), unless in remission from 5 years or more and judged of negligible potential of relapse
5. Known central nervous system metastases
6. Active viral hepatitis or chronic liver disease
7. Unstable cardiac condition, including congestive heart failure or angina pectoris, myocardial infarction within six months before enrollment, uncontrolled arterial hypertension or arrhythmia
8. Active major infection
9. Previous treatment with any other investigational or not investigational agents within 14 days of first day of study drug dosing
10. Known history of human immunodeficiency virus infection
11. Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation of the study drugs
12. Other serious concomitant illnesses or any condition that may interfere with the subject's participation in the study or evaluation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-28 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Time secondary resistance to Trabectedin | Week 18
  Time secondary resistance to Trabectedin is the time from the first trabectedin dose to progression not amenable to treatment with Trabectedin, or death, whichever occurs first

SECONDARY OUTCOMES:
Overall Survival | month 6,month 12, month 18, month 24, months 30, month 36, month 42, month 48, month 54, month 60
  Overall Survival is the time from the first trabectedin dose to death for any cause
Incidence of adverse event | Week 9, week 18, week 27, week 36, week 45, week 54, week 63, week 72, week 81
  Adverse events are evaluate from the first trabectedin dose throughout the study according to CTCAE 5.0
Progression free survival | Week 9, week 18, week 27, week 36, week 45, week 54, week 63, week 72, week 81
  Time from the first trabectedin dose to time of onset of progression disease

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Sanfilippo, MD, Principal Investigator — Fondazione IRCCS INT di Milano
Locations (15):
- Italy (15):
  - A.O. SS Antonio e Biagio e Cesare Arrigo, Alessandria, AL
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori - IRST, Meldola, FC
  - Istituto Europeo di Oncologia, Milan, MI
  - Istituto Clinico Humanitas, Rozzano, MI
  - Centro di Riferimento Oncologico di Aviano, Aviano, PD
  - Policlinico Universitario Campus Biomedico, Roma, RM
  - Fondazione del Piemonte per l'Oncologia IRCC Candiolo, Candiolo, Torino
  - Ospedale Gradenigo, Torino, TO
  - Istituto Ortopedico Rizzoli - Unit of Chemotherapy of Muscoloskeletal Tumors, Bologna
  - Azienda ospedaliero Universitaria Careggi di Firenze, Florence
  - Fondazione IRCCS INT Milano, Milan
  - Policlinico Federico II, Napoli
  - Irccs Istituto Oncologico Veneto (Iov), Padua
  - Ospedale Giaccone, Palermo
  - Istituti Fisioterapici Ospitalieri di Roma, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] D'Incalci M, Galmarini CM. A review of trabectedin (ET-743): a unique mechanism of action. Mol Cancer Ther. 2010 Aug;9(8):2157-63. doi: 10.1158/1535-7163.MCT-10-0263. Epub 2010 Jul 20. PMID 20647340
- [Background] Demetri GD, von Mehren M, Jones RL, Hensley ML, Schuetze SM, Staddon A, Milhem M, Elias A, Ganjoo K, Tawbi H, Van Tine BA, Spira A, Dean A, Khokhar NZ, Park YC, Knoblauch RE, Parekh TV, Maki RG, Patel SR. Efficacy and Safety of Trabectedin or Dacarbazine for Metastatic Liposarcoma or Leiomyosarcoma After Failure of Conventional Chemotherapy: Results of a Phase III Randomized Multicenter Clinical Trial. J Clin Oncol. 2016 Mar 10;34(8):786-93. doi: 10.1200/JCO.2015.62.4734. Epub 2015 Sep 14. PMID 26371143
- [Background] Sanfilippo R, Dileo P, Blay JY, Constantinidou A, Le Cesne A, Benson C, Vizzini L, Contu M, Baldi GG, Dei Tos AP, Casali PG. Trabectedin in advanced synovial sarcomas: a multicenter retrospective study from four European institutions and the Italian Rare Cancer Network. Anticancer Drugs. 2015 Jul;26(6):678-81. doi: 10.1097/CAD.0000000000000228. PMID 25763543
- [Background] Grosso F, Dileo P, Sanfilippo R, Stacchiotti S, Bertulli R, Piovesan C, Jimeno J, D'Incalci M, Gescher A, Casali PG. Steroid premedication markedly reduces liver and bone marrow toxicity of trabectedin in advanced sarcoma. Eur J Cancer. 2006 Jul;42(10):1484-90. doi: 10.1016/j.ejca.2006.02.010. Epub 2006 Jun 5. PMID 16737808
- [Background] Le Cesne A, Blay JY, Domont J, Tresch-Bruneel E, Chevreau C, Bertucci F, Delcambre C, Saada-Bouzid E, Piperno-Neumann S, Bay JO, Mir O, Ray-Coquard I, Ryckewaert T, Valentin T, Isambert N, Italiano A, Clisant S, Penel N. Interruption versus continuation of trabectedin in patients with soft-tissue sarcoma (T-DIS): a randomised phase 2 trial. Lancet Oncol. 2015 Mar;16(3):312-9. doi: 10.1016/S1470-2045(15)70031-8. Epub 2015 Feb 11. PMID 25680558